CLINICAL TRIAL: NCT02701075
Title: MC5-A Scrambler Therapy for the Treatment of Chronic Neuropathic Extremity Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Brooke Army Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Ann Marie Nayback-Beebe, PhD, RN, LTC Ann Marie Nayback-Beebe, Brooke Army Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TSNRP-N13-04
Record Dates: First submitted 2014-01-22; First posted 2016-03-08 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2017-02

CONDITIONS: Peripheral Neuropathy; Low Back Pain
Keywords: peripheral neuropathy; traumatic tissue injury; radiculopathy
MeSH Terms: conditions — Peripheral Nervous System Diseases; Low Back Pain; Radiculopathy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- MC5-A Scrambler Therapy (Experimental): MC5-A Scrambler Therapy is an electroanalgesia device that interferes with pain signal transmission by using nerve fibers as a passive means to convey a no pain message to the central nervous system. Electrodes are placed on dermatomes that correspond to the area of pain. Patient is treated for 30 minutes and given up to 10 treatment sessions.
  Interventions: Device: MC5-A Scrambler Therapy
- MC5-A Scrambler Therapy Sham Device (Sham Comparator): The MC5-A Scrambler Therapy Device will be used as an active sham device in this randomized double blind study. Participants assigned to this arm will not receive active therapy.
  Interventions: Device: MC5-A Scrambler Therapy Sham Device

INTERVENTIONS:
Device: MC5-A Scrambler Therapy — up to 10 sessions, each session lasting 30 minutes
  Other Names: Calmare
  Arms: MC5-A Scrambler Therapy
Device: MC5-A Scrambler Therapy Sham Device — up to 10 sessions, each session lasting 30 minutes
  Other Names: Calmare Sham
  Arms: MC5-A Scrambler Therapy Sham Device

SUMMARY:
The FDA-approved MC5-A Scrambler Therapy (MC5-A ST) is an electroanalgesia device that interferes with pain signal transmission by using nerve fibers as a passive means to convey a message of normality (sans pain) to the central nervous system. While preliminary research has demonstrated its efficacy in treating chronic neuropathic pain secondary to cancer and failed back surgery syndrome, its effectiveness in treating chronic neuropathic pain secondary to traumatic musculoskeletal injuries like those experienced in combat has not been investigated. The purpose of this prospective, double-blind, randomized controlled, study is to determine if the MC5-A ST is efficacious in altering the biological, psychological, and social components of the chronic neuropathic pain experience in military Service Members (SMs) with traumatic musculoskeletal extremity injuries.

ELIGIBILITY:
Inclusion Criteria:

* military service members (active duty & retirees) between the ages of 18 and 79, inclusive
* neuropathic pain symptoms present for 3 months or greater prior to entry into the study
* rated pain intensity equal to or greater than 3 on NRS-11 pain scale
* painful peripheral neuropathy in an extremity that is the result of a traumatic injury (post-traumatic/ post-surgical neuropathy, stump pain, entrapment neuropathy), or low back pain with radiculopathy
* stable pain medication treatment regimen
* able to speak and read English, understand the study procedures, and consent to study participation

Exclusion Criteria:

* pacemaker or other implantable devices
* vena cava, aneurysm clips, coronary or other vascular stents
* pregnancy via a pregnancy test
* history of epilepsy, brain injury, symptomatic brain metastases
* prior celiac plexus block, or other neurolytic pain control treatment, within 4 weeks
* wounds or skin irritation in areas where the electrodes are required to be placed
* cardiac ischemia within the previous 6 months
* severe arrhythmia
* documented history of moderate or severe traumatic brain injury
* latex allergies
* open wound over site of chronic pain
* unable to stop anti-epileptic medications or gabapentin over 2 weeks of MC5-A ST treatment
* history of electroanalgesia treatment (electroacupuncture, biomodulator, TENS) over last 30 days
* participation in the study would delay the medical board (MEB) processing of the service member off of active duty status or would delay a return to duty status to their home unit.
* metal implants such as cardiac pacemakers, automatic defibrillators, aneurysm clips, vena cava clips and skull plates

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2013-09; Primary Completion 2016-12 (Actual); Study Completion 2017-08-31 (Estimated)

PRIMARY OUTCOMES:
Change over time in pain on the Numerical Rating Scale-11 Pain Score (NRS-11) | Baseline, Week 3, Week 6

SECONDARY OUTCOMES:
Change over time in oral consumption of analgesic medications | Baseline, Week 3, Week 6

OTHER OUTCOMES:
Change over time in depressive symptoms on the Patient Health Questionnaire-9 (PHQ-9) at week 3 | Baseline, Week 3, Week 6
Change over time in anxiety symptoms on the Generalized Anxiety Disorder-7 (GAD-7) | Baseline, Week 3, Week 6
Change over time in posttraumatic stress symptoms on the Posttraumatic Stress Disorder Checklist - Military (PCL-M) | Baseline, Week 3, Week 6
Change over time in quality of sleep symptoms on the Pittsburgh Quality of Sleep Index (PQSI) | Baseline, Week 3, Week 6
Change over time in perception of health on the Quality Of Life - Health Survey (SF-12) | Baseline, Week 3, Week 6
Change over time in the perception of social support on the Interpersonal Relationships Inventory Short Form (IPRI-SF) | Baseline, Week 3, Week 6
Abbreviated Acceptability Rating Profile | Week 6

CONTACTS AND LOCATIONS:
Overall Officials: Ann Marie Nayback-Beebe, PhD, FNP-BC, Principal Investigator — Brooke Army Medical Center
Locations (1):
- Brooke Army Medical Center, Fort Sam Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No